CLINICAL TRIAL: NCT05983224
Title: Effect of Quercetin Supplementation on Glycemic Status, Lipid Profile, Oxidative Stress, Inflammation, Growth Factor, Adiponectin, Sex Hormones and Anthropometric Indices in Women With Endometriosis
Brief Title: Effect of Quercetin Supplementation on Endometriosis Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ghazaleh Eslamian, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 43003154
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Endometriosis
Keywords: Quercetin; Endometriosis; Inflammation; Gonadal Steroid Hormones; Anthropometric; Adiponectin; Growth factor; Metabolic factors
MeSH Terms: conditions — Endometriosis; Inflammation | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quercetin (Experimental): The intervention group will receive two 500 mg quercetin tablets daily, after breakfast and lunch, for twelve weeks.
  Interventions: Dietary Supplement: Quercetin
- Placebo (Placebo Comparator): The Placebogroup will receive Placebo tablets daily, after breakfast and lunch, for twelve weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Quercetin — The intervention group will receive two 500 mg quercetin tablets daily, after breakfast and lunch, for twelve weeks.
  Arms: Quercetin
Other: Placebo — The control group will receive two placebo daily, after breakfast and lunch, for twelve weeks.
  Arms: Placebo

SUMMARY:
Quercetin is a polyphenol compound that possesses anti-inflammatory properties and can be found in various food sources like apples, berries, cabbage, and onions. In Park et al.'s study, it was discovered that quercetin led to a significant decrease in the proliferation of endometriosis cells. Furthermore, quercetin also triggered apoptosis in endometriosis cells in vitro and reduced the size of endometriosis lesions in vivo. Nevertheless, as of now, there have been no studies conducted in Iran or worldwide that explore the effects of quercetin supplementation on individuals with endometriosis. Hence, the aim of this study is to investigate the impact of quercetin supplementation on factors such as glycemic status, lipid profile, oxidative stress, inflammation, growth factors, adiponectin, sex hormones, and anthropometric indicators in women suffering from endometriosis.

DETAILED DESCRIPTION:
The participants in the study were randomly assigned to two groups: the intervention group and the control group. The intervention group will receive two 500 mg quercetin tablets daily, after breakfast and lunch, for twelve weeks. On the other hand, the control group will be given a placebo. Blood samples will be collected before and after the intervention to measure changes in blood lipid profile, fasting blood sugar, sex hormones (testosterone, estrogen, progesterone), TNFα, IL-6, adiponectin, IGF1, HbA1C, SHBG, FSH, LH, and plasma total antioxidant capacity.

ELIGIBILITY:
Inclusion Criteria:

* Willing to cooperate and complete the informed consent form.
* Diagnosed endometriosis using laparoscopy and histopathological tests.
* In the age group of 18 to 40 years.
* Having a regular menstrual cycle.
* Having a body mass index between 18.5 and 30.

Exclusion Criteria:

* Using hormonal medications or intrauterine treatments for a minimum of three months prior to collecting a sample.
* Having immune system disorders, persistent infections, diabetes, or any conditions like polyps and fibroids within the uterine cavity.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean serum TNF-alpha concentration | 12 weeks
  Human Tumor Necrosis Factor Αlpha, TNF-A ELISA Kit
Mean serum IL-6 concentration | 12 weeks
  Human Interleukin 6, IL-6 ELISA Kit

SECONDARY OUTCOMES:
Mean Serum FBS concentration | 12 weeks
  Glucose Test Kit
Mean HbA1C Serum | 12 weeks
  Human Hemoglobin A1c (HbA1c) Assay Kit
Mean Serum Testosterone concentration | 12 weeks
  The Testosterone ELISA Kits
Mean Serum Estrogen concentration | 12 weeks
  The Total Estrogens ELISA Assay Kit
Mean Serum Adiponectin concentration | 12 weeks
  Adiponectin Human ELISA Kit
Mean Serum IGF1 concentration | 12 weeks
  IGF-1 ELISA Assay Kit
Mean Serum SHBG concentration | 12 weeks
  liquid chromatography-tandem mass spectrometry
Mean Serum FSH concentration | 12 weeks
  FSH (Human) ELISA Kit
Mean Serum LH concentration | 12 weeks
  LH (Human) ELISA Kit
Mean Serum Progesterone concentration | 12 weeks
  The Progesterone Enzyme Immunoassay Kit
Mean plasma total antioxidant capacity concentration | 12 weeks
  Total Antioxidant Capacity ELISA Kit

CONTACTS AND LOCATIONS:
Overall Officials: Ghazaleh Eslamian, PhD, Principal Investigator — National Nutrition and Food Technology Research Institute
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after starting the study

REFERENCES:
- [Background] Khorshidi M, Moini A, Alipoor E, Rezvan N, Gorgani-Firuzjaee S, Yaseri M, Hosseinzadeh-Attar MJ. The effects of quercetin supplementation on metabolic and hormonal parameters as well as plasma concentration and gene expression of resistin in overweight or obese women with polycystic ovary syndrome. Phytother Res. 2018 Nov;32(11):2282-2289. doi: 10.1002/ptr.6166. Epub 2018 Jul 30. PMID 30062709
- [Background] Rezvan N, Moini A, Gorgani-Firuzjaee S, Hosseinzadeh-Attar MJ. Oral Quercetin Supplementation Enhances Adiponectin Receptor Transcript Expression in Polycystic Ovary Syndrome Patients: A Randomized Placebo-Controlled Double-Blind Clinical Trial. Cell J. 2018 Jan;19(4):627-633. doi: 10.22074/cellj.2018.4577. Epub 2017 Nov 4. PMID 29105398